CLINICAL TRIAL: NCT00266461
Title: A Randomized, Controlled, Open-Label Tolerability And Efficacy Study Of TU-100 For The Treatment Of Postoperative Ileus In Patients Undergoing Laparotomy For Large Bowel Resection
Brief Title: A Tolerability and Efficacy Study of TU-100 For The Treatment of Postoperative Ileus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TU100P2T1
Record Dates: First submitted 2005-12-14; First posted 2005-12-16 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Postoperative Ileus
Keywords: Postoperative Ileus
MeSH Terms: interventions — 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TU-100 7.5g/day (Experimental): Subjects will be randomized to TU-100 7.5g, 15g, or no active treatment group. Subjects will take a daily dose divided into 3 times a day.
  Interventions: Drug: Daikenchuto Extract Granules (TU-100)
- TU-100 15g/day (Experimental): Subjects will be randomized to TU-100 7.5g, 15g, or no active treatment group. Subjects will take a daily dose divided into 3 times a day.
  Interventions: Drug: Daikenchuto Extract Granules (TU-100)
- Water (No Intervention): Subjects will be randomized to TU-100 7.5g, 15g, or no active treatment group. Subjects will take a daily dose divided into 3 times a day.

INTERVENTIONS:
Drug: Daikenchuto Extract Granules (TU-100)
  Arms: TU-100 15g/day; TU-100 7.5g/day

SUMMARY:
Postoperative ileus (POI), a transient impairment of gastrointestinal (GI) motility, commonly occurs in patients who have undergone abdominal surgery and contributes to postoperative morbidity, including delayed enteral nutrition, increased patient discomfort, and prolonged hospitalization. POI appears to be have many causes, with activation of inhibitory reflexes, inflammatory responses, and the effects of anesthesia and analgesics all playing roles. However, there is no approved pharmacological therapy for the treatment and prevention of POI.

Daikenchuto (TU-100) is an herbal formulation consisting of Asian ginseng, Zanthoxylum fruit (Sichuan pepper), ginger, and malt sugar, which was originally described in Jin kui yao lue, the classical medical textbook written in ancient China in the third century by Zhang Zhong Jing. Since it was introduced to Japan, Daikenchuto has been used in the treatment of abdominal pain and a feeling of coldness in the abdomen.

TSUMURA Daikenchuto Extract Granules, Product Code TU-100, is a modern herbal product manufactured in the dosage form of granules by Tsumura & Co. The current Tsumura product, TU-100, was approved for manufacture as a prescription drug in 1986 by the Japanese Ministry of Health and Welfare and has been sold commercially as a prescription Kampo (a generic term for the system of traditional medicine that was developed in Japan after being introduced from China in the fourth century) drug in Japan for many years. The drug product proposed for use in the clinical studies is identical to the drug currently sold in Japan. In addition, all three botanical components and maltose syrup powder are considered as food substances and are currently part of the United States food supply.

The purpose of this study evaluate the tolerability, efficacy and safety of TU-100 for the treatment of postoperative ileus (POI) in patients undergoing laparotomy for large bowel resection

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label study designed to evaluate the tolerability and efficacy of TU-100 for the treatment of POI in patients undergoing laparotomy for large bowel resection. It will be conducted at multiple centers in the United States. A total of 24 patients will be enrolled in the study. Patient participation in the study will last for up to 32 days (from Screening to postoperative day 10 [POD 10] or until the time when a discharge order is written for the patient, whichever comes first), with follow-up safety assessments to occur 7 and 14 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a patient must meet all of the following criteria:

1. Is at least 18 years of age;
2. Is male or female. Female patients cannot be pregnant or lactating and must be surgically sterile, postmenopausal (no menses for the previous 12 months), or practicing an effective method of birth control as determined by the investigator (eg, oral contraceptives, double barrier methods, hormonal injectable or implantable contraceptives, tubal ligation, or partner with vasectomy);
3. Has been diagnosed with sigmoid carcinoma; ascending, transverse, or descending colon carcinoma; colonic polyps; carcinoid tumors; lymphoma localized to the abdomen; ischemic bowel; toxic megacolon with no perforation; any tumor of the bowel determined to require removal; or diverticulitis;
4. Requires laparotomy for large bowel resection. Note: patients who are shifted to laparotomy during laparoscopic surgery are acceptable;
5. Is hospitalized for surgery and recovery;
6. Has a pre-operative Karnofsky performance status of 80% to 100%; and
7. Provides written informed consent prior to participation in the study after full explanations of the study purpose and procedures.

Exclusion Criteria:

In order to participate in this study, a patient must not meet any of the following criteria:

1. Has been diagnosed with Crohn's disease, ulcerative colitis, or irritable bowel syndrome. Note: patients with inactive ulcerative colitis who are in stable clinical remission and/or on maintenance therapy to prevent relapse are acceptable;
2. Is a pregnant or lactating female;
3. Requires a colostomy or any other ostomy device placement;
4. Requires emergency surgery or has surgery in the presence of an ongoing infection, including bowel obstruction and perforated bowel;
5. Has colorectal cancer with a Dukes Classification score of D;
6. Has diabetic neuropathy;
7. Has a history of gastroparesis;
8. Has a compromised immune system, either from treatment with corticosteroids or other immunosuppressive agents within 2 weeks of surgery or from immunosuppressive diseases (eg, human immunodeficiency virus); Note: patients on chronic treatment (for at least 3 months) with corticosteroids of up to 10 mg daily of prednisone or equivalent are acceptable if dosing has been stable for at least 2 weeks;
9. Has any other serious condition that might adversely affect their safety or ability to participate in this study, such as liver disorders (including alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] levels greater than 2.5 times the upper limit of normal [ULN]), kidney disorders, heart failure, blood disorders, or metabolic disorders;
10. Has a history of any allergic reactions to ginseng, ginger, Zanthoxylum fruit (Sichuan pepper), or maltose;
11. Has a history of narcotic drug abuse (especially heroin or opium) or chronic narcotic use for pain management within 2 weeks of surgery;
12. Requires anticancer radiation or chemotherapy within 2 weeks of surgery;
13. Has a history of laparotomy or laparoscopy other than simple laparoscopic procedures such as cholecystectomy, gynecological procedures, or inguinal hernia repair. Note: a history of laparoscopic fundoplication is exclusive, while a history of appendectomy or hysterectomy is acceptable; patients who have had laparotomy procedures in the past with no history of subsequent small bowel or large bowel obstruction are acceptable;
14. Has a history of any type of ileus;
15. Has a history of receiving abdominal radiation therapy in addition to subsequent small bowel or large bowel obstruction. Note: a history of radiation therapy with no small bowel or large bowel obstruction is acceptable; a history of pelvic radiation therapy is also acceptable;
16. Is unwilling or unable to comply with the procedures described in this protocol or is otherwise unacceptable for enrollment in the opinion of the investigator; and
17. Has participated in any other investigational product or device trial within 30 days prior to enrolling in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the tolerability of TU-100 for the treatment of postoperative ileus (POI) in patients undergoing laparotomy for large bowel resection based on the incidence of adverse events (AEs). | Up to 10 days

SECONDARY OUTCOMES:
To evaluate the safety of TU-100 in the treatment of POI based on an assessment of objective and subjective symptoms and clinical laboratory data | Up to 10 days
To evaluate the efficacy of TU-100 in the treatment of POI based on the length of time from the end of surgery to gastrointestinal(GI) function recovery and time to discharge order, and | Up to 10 days
To determine the acceptability of TU-100 to American patients based on the number of discontinuations due to noncompliance and an assessment of taste. | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Shunji Mochida, PhD, Study Director — Tsumura USA Inc.
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States